CLINICAL TRIAL: NCT02391649
Title: A Randomized Controlled Trial of Problem-solving Based Bibliotherapy Program for Family Caregivers of People With Psychotic Disorders
Brief Title: Problem-solving-based Bibliotherapy Program for Family Caregivers
Acronym: PSBBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Castle Peak Hospital (Other Government); Prince of Wales Hospital, Shatin, Hong Kong (Other); University of Victoria (Other)
Responsible Party: Principal Investigator, Prof. Wai Tong CHIEN, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 15401114
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: psychosis; self-learning program; problem-solving; family caregivers; randomized controlled trial
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Repeated-measures, three-arm design (and in phase 1, two pilot 2-arm controlled trials with repeated-measures design; sample size 112 for the two pilot studies)
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blind to the group assignment and intervention undertaken and concealed to the participant list.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Self-learning program (Experimental): The participants in the Problem-solving Based Self-learning Program will complete the self-help and problem-solving manual developed by the research team for caregivers of people with psychotic disorders over 20 weeks. In addition to the orientation, understanding about psychosis and its care and final review sessions (4 sessions in 3 weeks) facilitated by the research nurse, the caregivers will work independently through the modules over 15-17 weeks.
  Interventions: Behavioral: Self-learning program
- Psycho-education (in Phase 2) (Active Comparator): Two trained advanced practice psychiatric nurses who are experienced in psychiatric rehabilitation and group programs will lead the psychoeducation group, which is guided by a validated treatment protocol based on the research team's and McFarlane and his colleagues' psychoeducation programs for psychosis. The program consists of 12 two-hour sessions held weekly/biweekly (similar to the self-learning program, completed in 5 months), with 4 main components, including 'introduction and goal setting'; 'an education workshop on mental illness, treatment and community services'; 'group exercises/rehearsals and discussion on symptom management, coping and self-care'; and ''review and future plan'.
  Interventions: Behavioral: Psycho-education program (in Phase 2)
- Routine community care (No Intervention): Participants in the control group (and treatment groups) will receive routine psychiatric outpatient and family services.

INTERVENTIONS:
Behavioral: Self-learning program — The PSBBP in this study consists of 5 modules (Module 1: Caregiver's well-being; Module 2:Getting the best out of support services; Module 3:Well-being of the person with schizophrenia; Module 4:Dealing with the [psychosocial] effects of the illness; and Module 5:Dealing with [physical and mental health] effects of the illness), helping each caregiver from developing a positive attitude to caregiving, identifying caring related problems and obstacles, predicting positive and negative implications of each alternative, to trying out the solution and monitor if it worked.
  Arms: Self-learning program
Behavioral: Psycho-education program (in Phase 2) — The program consists of 12 two-hour sessions held weekly/biweekly completed in 5 months, with 4 main components, including 'introduction and goal setting'; 'an education workshop on mental illness, treatment and community services'; 'group exercises/rehearsals and discussion on symptom management, coping and self-care'; and 'review and future plan'.
  Arms: Psycho-education (in Phase 2)

SUMMARY:
This proposed randomized controlled trial will test the effectiveness of a problem-solving based bibliotherapy program (PSBBP) for Chinese family caregivers in psychotic disorders (not more than 5 years onset). A repeated-measures, three-group design will be used to evaluate and compare the effects between two treatment groups(PSBBP and psycho-education group) and routine outpatient service and family support (control group) for 198 randomly selected family caregivers of outpatients with psychotic disorders over a 24-month follow-up.

Before the 3-arm trial to be conducted, a pilot parallel-group randomised controlled trial with a similar study design to the later three-arm randomised controlled trial (Phase 2) will be conducted at one psychiatric outpatient clinic in Hong Kong. Receiving an additional funding from local government, another pilot two-arm trial will also be conducted for family caregivers of people with first-episode psychosis in the community to support and inform the 3-arm randomised controlled trial.

DETAILED DESCRIPTION:
Family caregivers of people with psychotic disorders are confronted by a various physical, psychosocial and financial hardships. This can adversely affect family members' caregiving experiences, psychological distress, general well-being, and family relationships or emotional involvement, which in turn may contribute to a greater risk of patient relapse and non-recovery. While family psycho-education and mutual support groups are effective in reducing caregivers' burden of care, these approaches usually require regular meetings and encounter difficulties in extensive training of group leaders/facilitators and engaging participants to actively share their caregiving experiences due to time inconvenience and fear/inability of expression of feelings. By virtue of the above, an alternate model of self-help program in book form named bibliotherapy, which is a guided reading and self-practice program with problem-solving training facilitated by a psychiatric nurse, has recently demonstrated evidences in clinical trials for families of depressive and psychotic patients by the research team, and other researchers.

In phase 1, a pilot randomised controlled trial with repeated measures, parallel-group (2-arm) design will be carried out at one psychiatric clinic. This pilot trial aims to evaluate the effects between the treatment group (i.e., a problem-solving based self-learning program) and routine outpatient service (control group) for 116 randomly selected family caregivers of outpatients with recent-onset psychosis over a 6-month follow-up. The study outcomes include the caregivers' burden of care, caregiving experiences, and problem-solving abilities, and the patients' mental state, functioning, and re-hospitalization rates. They will be measured at recruitment, one week, and 6 months following the interventions.

Another pilot controlled trial will recruit 116 families of people with first-episode psychosis attending follow-up at two regional psychiatric outpatient clinics in Hong Kong. Participant will be randomly selected in equal proportion from the two clinics under study and after baseline measures, the participants will be randomised to the treatment (i.e., the Chinese version of the original manual of bibliotherapy program) or the routine care. They will also be measured with the similar outcomes at the above pilot study at recruitment, one week, 6 months, and 12 months post-intervention.

In phase 2, a 3-arm randomized controlled trial will be conducted to test the effectiveness of the problem-solving based bibliotherapy program (PSBBP) for Chinese family caregivers in early stage of psychotic disorders. A repeated-measures, three-group design will be used to evaluate and compare the effects between two treatment groups (PSBBP and psycho-education group) and routine outpatient service and family support (control group) for 198 randomly selected family caregivers of outpatients with psychotic disorders over a 24-month follow-up. Primary outcomes include caregivers' burden of care, caregiving experiences and coping and social problem-solving skills using validated instruments. Secondary outcomes are patients' mental state, functioning, perceived expressed emotion, and re-hospitalization rate. They will be measured at recruitment, one week, and 12 and 24 months following the interventions. It is hypothesized that the PSBBP participants will produce significantly better improvements in caregivers' perceived burden, caregiving experience and coping and problem-solving skills than those in psycho-education and control groups over 24-month follow-up.

Focus group interviews will be conducted after the first post-test with 20 caregivers (10 participants per group) in both treatment groups. Their data will be content analyzed to identify their perceived benefits, limitations and difficulties encountered and therapeutic ingredients of the two programs.

ELIGIBILITY:
Inclusion Criteria of the participants include those who:

* Hong Kong Chinese residents, aged 18-60;
* taking care of and living with a family member primarily diagnosed with one psychotic disorder in the past 5 years (for Phase 1, patients with recent-onset [12 months] or first-episode psychosis will be recruited);
* able to read and understand Cantonese/Mandarin; and
* perceived a moderate to high burden of care (measured by Family Burden Interview Schedule (>20 out of 50 scores)

Exclusion criteria of family caregivers include:

* those received or are receiving another family intervention;
* those are having cognitive impairment or learning disability; and/or
* those presented with a recent personal history of a serious mental illness or medical disease that may adversely affect their ability to participate in the intervention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 422 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Perceived burden of care (Chinese version of the 25-item Family Burden Interview Schedule) | 6 months (for Phases 1 and 2) after completion of intervention
  Caregivers' perceived burden of care will be measured by a Chinese version of the 25-item Family Burden Interview Schedule.
Perceived burden of care (Chinese version of the 25-item Family Burden Interview Schedule) | 12 months (for Phases 1 and 2) after completion of intervention
  Caregivers' perceived burden of care will be measured by a Chinese version of the 25-item Family Burden Interview Schedule.
Perceived burden of care (Chinese version of the 25-item Family Burden Interview Schedule) | 24 months (for Phase 2 only) after completion of intervention
  Caregivers' perceived burden of care will be measured by a Chinese version of the 25-item Family Burden Interview Schedule.
Coping style (42-item Revised Ways of Coping Checklist) | 6 months (for Phases 1 and 2) after completion of intervention
  A Chinese version of Coping style of the caregivers style will be assessed using the 42-item Revised Ways of Coping Checklist.
Coping style (42-item Revised Ways of Coping Checklist) | 12 months (for Phases 1 and 2) after completion of intervention
  A Chinese version of Coping style of the caregivers style will be assessed using the 42-item Revised Ways of Coping Checklist.
Coping style (42-item Revised Ways of Coping Checklist) | 24 months (for Phase 2 only) after completion of intervention
  A Chinese version of Coping style of the caregivers style will be assessed using the 42-item Revised Ways of Coping Checklist.

SECONDARY OUTCOMES:
Experience of caregiving (Chinese version of Experience of Caregiving Inventory) | 24 months (Phase 2; 6 and 12 months for Phase 1) after completion of intervention
  The Chinese version of Experience of Caregiving Inventory is a 66-item self-reporting scale that measures experiences of caregiving to a family member with mental illness based on the transactional model of stress-appraisal-coping.
Social Problem-Solving (Chinese version of Revised (Short) Social Problem-Solving Inventory) | 24 months (Phase 2; 6 and 12 months for Phase 1) after completion of intervention
  The Chinese version of Revised (Short) Social Problem-Solving Inventory will be used to assess participants' problem solving.
Mental state (Positive and Negative Syndrome Scale) | 24 months (Phase 2; 6 and 12 months for Phase 1) after completion of intervention
  Patients' mental state will be evaluated by the Positive and Negative Syndrome Scale, a 30-item inventory assessing the absence/severity of psychotic symptoms across positive symptoms, negative symptoms and general psycho-pathology symptoms.
Patient functioning (43-item Specific Level of Functioning Scale) | 24 months (Phase 2; 6 and 12 months for Phase 1) after completion of intervention
  The 43-item Specific Level of Functioning Scale will be used to assess 3 functional domains for patients with schizophrenia spectrum disorders, including physical functioning/personal care (12 items), social functioning (14 items) and community living skills (17 items) on a 5-point Likert scale.
Perceived expressed emotion (Level of Expressed Emotion scale; used in Phase 2 only) | 24 months after completion of intervention
  Perceived expressed emotion by patients will be measured by Level of Expressed Emotion scale.The scale comprises 4 domains: intrusiveness, attitude toward illness, tolerance/expectancy, and emotional responses; each consists of 15 items on a 4-point Likert scale ('1-Not true' to '4-True').
Rate and length of re-hospitalizations | 24 months (Phase 1; 6 and 12 months for Phase 1) after completion of intervention
  The data of patients' frequency and lengths (days) of psychiatric hospitalizations over the intervention period, 6 months, 12 months or 24 months follow-ups, will be recorded by the research assistant by reviewing the electronic patient records.

CONTACTS AND LOCATIONS:
Overall Officials: Wai Tong CHIEN, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - Li Ka Shing Specialty OPD, Shatin, NT
  - TM Psy Centre, Tuenmen, NT

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chien WT, Chan SW. Testing the psychometric properties of a Chinese version of the Level of Expressed Emotion scale. Res Nurs Health. 2009 Feb;32(1):59-70. doi: 10.1002/nur.20303. PMID 18800379
- [Background] McCann TV, Lubman DI, Cotton SM, Murphy B, Crisp K, Catania L, Marck C, Gleeson JF. A randomized controlled trial of bibliotherapy for carers of young people with first-episode psychosis. Schizophr Bull. 2013 Nov;39(6):1307-17. doi: 10.1093/schbul/sbs121. Epub 2012 Nov 20. PMID 23172001
- [Background] Chien WT, Lee IY. The schizophrenia care management program for family caregivers of Chinese patients with schizophrenia. Psychiatr Serv. 2010 Mar;61(3):317-20. doi: 10.1176/ps.2010.61.3.317. PMID 20194413
- [Background] Chien WT, Leung SF, Yeung FK, Wong WK. Current approaches to treatments for schizophrenia spectrum disorders, part II: psychosocial interventions and patient-focused perspectives in psychiatric care. Neuropsychiatr Dis Treat. 2013;9:1463-81. doi: 10.2147/NDT.S49263. Epub 2013 Sep 25. PMID 24109184
- [Background] Breitborde NJ, Moreno FA, Mai-Dixon N, Peterson R, Durst L, Bernstein B, Byreddy S, McFarlane WR. Multifamily group psychoeducation and cognitive remediation for first-episode psychosis: a randomized controlled trial. BMC Psychiatry. 2011 Jan 12;11:9. doi: 10.1186/1471-244X-11-9. PMID 21226941
- [Result] Chien WT, Yip AL, Liu JY, McMaster TW. The effectiveness of manual-guided, problem-solving-based self-learning programme for family caregivers of people with recent-onset psychosis: A randomised controlled trial with 6-month follow-up. Int J Nurs Stud. 2016 Jul;59:141-55. doi: 10.1016/j.ijnurstu.2016.03.018. Epub 2016 Apr 6. PMID 27222459